CLINICAL TRIAL: NCT03378024
Title: To Evaluate the Correlation of Near Infrared Spectroscopy, ABI, Exercise Test, baPWV and Microalbuminuria With Peripheral Artery Occlusion Disease and Other Atherosclerosis Outcome
Brief Title: Evaluate the Correlation of NIRS, ABI, Exercise, baPWV and Albuminuria With Peripheral Artery Occlusion Disease (PAD) and Other Atherosclerosis Outcomes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG2F0181
Record Dates: First submitted 2017-05-04; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Peripheral Arterial Occlusive Disease
Keywords: Oscillometric device; repetitive Active Pedal Plantarflexion (APP) exercise test; brachial-ankle pulse wave velocity (baPWV)
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Arterial Occlusive Disease 1; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- diabetic mellitus patients: Measure the brachial-ankle pulse wave velocity (baPWV) and the resting ankle-brachial index(ABI) of pre-exercise and post-exercise by the oscillometric (Omron Colin co.).
  And follow up for 3 years to identify of the correlation with PAD outcome.
  Interventions: Device: oscillometric (Omron Colin co)

INTERVENTIONS:
Device: oscillometric (Omron Colin co) — fast measurements of the brachial-ankle pulse wave velocity (baPWV) and the resting ankle-brachial index(ABI) with the oscillometric method (Omron Colin co, Japan)

SUMMARY:
By utilizing Near infrared spectroscopy (NIRS), the local blood flow, tissue oxygenation (StO2), and recovery time of ischemic leg; can be determined. It is reasonable to standardize an easy, simple and safe Active Pedal Plantarflexion (APP) exercise test working load which can achieve the lowest StO2 and other parameters in ischemic leg through observation of NIRS. After standardized of an effective APP test, a determination of a new cutoff value of resting ABI in diagnosing PAD can probably be searched. Analysing the correlation of baPWV with ABI, atherosclerosis risk factors and parameters with atherosclerosis outcome. Observation the Sequential changes of baPWV, ABI and microalbuminuria after managing the atherosclerosis risks, and analyze their influence on the outcome of PAD, coronary artery disease(CAD) and cerebral vascular disease(CVA) outcomes.

DETAILED DESCRIPTION:
Exercise testing by Active Pedal Plantar flexion:

The investigators plan to collect 140 cases:

1. Healthy subjects with no apparent atherosclerotic risk [< 65 y/o, no diabetic mellitus (DM), no hypertension, or no hyperlipidemia, not obese, not current smoker, no smoking history >10 years] 4(n=5)
2. Patients at risks (e.g. hypertension, hyperlipidemia) (n=5) but without DM,
3. Type 1 and Type 2 DM patients with normal ABI( >1.0)and normal Toe-brachial index (TBI) (> 0.6) without intermittent claudication(by Edinburgh claudication questionnaire), nor PAD diagnosis (n= 10)
4. DM normal ABI>1.0 and normal TBI (> 0.6) with suspected symptoms (intermittent claudication, non healing ulcer) (n=10),
5. DM normal or borderline ABI( >1, 0.91~0.99) but low TBI (< 0.6), or with suspected symptoms (intermittent claudication, non healing ulcer) (n=20),
6. DM patients with borderline ABI (0.91-0.99) (n=50) with or without leg symptoms,
7. DM patients abnormal Low ABI (<0.9) (n=30) with or without leg symptoms,
8. DM patients abnormal high ABI (> 1.3) (n=10)with or without leg symptoms, Post-exercise ABI with APP, and NIRS examination during APP exercise test will be performed.

The investigators also plan to collect 500 cases of nonpregnant, ≥ 40 years old DM patients, obtained baPWV and the resting ABI by oscillometric device (Omron colin, Japan). The investigators will apply this novel technique to assess the extent of arteriosclerosis and atherosclerosis by oscillometric device in our DM patient without PAD (ABI >0.9).

Collect baseline characteristics and follow up annual data: Age, sex, body weight, height, BMI, waist circumferences, history of smoking (ex-smoker, current), coexisting hypertension, hyperlipidemia, DM duration, presence of chronic DM complications of neuropathy, retinopathy (by fundus camera), nephropathy (cr, estimate glomerular filtration rate(eGFR), proteinuria, microalbuminuria). The biochemistry data involving atherosclerotic risk including: systolic blood pressure, diastolic pressure, mean pulse pressure, HbA1c, total cholesterol, LDL-Cholesterol(LDL-C), HDL-Cholesterol(HDL-C), triglyceride, creatinine, microalbuminuria,, high sensitive C-Reactive Protein (hs CRP), baseline EKG all will be collected. All the above data will be followed up annually for 3 years to analyze the correlation of progressive change of baPWV, ABI and microalbuminuria with the atherosclerosis event and mortality.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetic patients
* type 2 diabetic patients

Exclusion Criteria:

* Pregnancy
* Critical limb ischemia (gangrene change)
* A permanent pacemaker implant
* Systolic BP ≥ 200 mmHg or diastolic BP ≥100 mmHg
* Symptomatic orthostatic blood pressure drop ≥ 20 mmHg
* Severe critical aortic stenosis
* Acute medical illness, fever, systemic infection
* Uncontrolled atrial or ventricular dysrhythmias
* Uncontrolled sinus tachycardia≥ 120/min
* Peripheral venous insufficiency, thrombosis or thrombophlebitis
* Those who has factors known to influence the PWV
* The brachial-ankle PWV could not be measured on the right and left sides
* Orthopedic condition (ankle or foot) that cannot perform an active pedal plantar flexion (APP) technique (arthritis, hemiparesis, balance impairment etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nonpregnant & ≥ 20 years old type1 and type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Define the correlation between NIRS and ABI | 12 month
  Analyse the correlation of NIRS with different ABI
Defined APP exercise ABI criteria for PAD diagnosis | 12 month
  Design APP exercise with effective working load to defined ABI criteria for PAD diagnosis
The correlation of changes of baPWV and the outcome of PAD | 12,24 and 36 months
  Analyse the sequential changes of baPWV and the outcome of PAD
The correlation of changes of exercise ABI and the outcome of PAD | 12,24 and 36 months
  Analyse the sequential changes of exercise ABI and the outcome of PAD
The correlation of changes of albuminuria and the outcome of PAD | 12,24 and 36 months
  Analyse the sequential changes of albuminuria and the outcome of PAD

CONTACTS AND LOCATIONS:
Overall Officials: Ng Soh Ching, MD, Principal Investigator — Chang Gung Memorial Hospital, Keelung

IPD SHARING:
Plan to Share IPD: No